CLINICAL TRIAL: NCT04913935
Title: Investigation of Parameters of Trapeziometacarpal Joint Configuration and Tenar Muscles in Patients With TMC OA
Brief Title: Investigation of Thenar Muscles Morphometric Parameters in Patients With TMC OA
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Feray Karademir, Research Asssistant, Hacettepe University
Other Study IDs: GO 18/204
Record Dates: First submitted 2019-08-08; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Thumb Osteoarthritis; Muscle Atrophy or Weakness
Keywords: thumb; trapeziometacarpal osteoarthritis; muscle thickness; muscle cross sectional area; hand function; hand dexterity; pain; pinch strength
MeSH Terms: conditions — Muscular Atrophy; Asthenia; Pain | interventions — Radiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TMC OA: women who were diagnosed with TMC OA
  Interventions: Diagnostic Test: Muscle-Skeleton Ultrasonography
- Control: healty volunteer women
  Interventions: Diagnostic Test: Muscle-Skeleton Ultrasonography

INTERVENTIONS:
Diagnostic Test: Muscle-Skeleton Ultrasonography — postero-anterior radiography
  Other Names: Radiography

SUMMARY:
In this study, investigators aimed to investigate the morphometric parameters tenar muscles and joint configuration in patients with trapeziometacarpal osteoarthritis (TMC OA) osteoarthritis stages, thenar muscle parameters, radial subluxation rate, functional level and hand dexterity.

DETAILED DESCRIPTION:
Patients diagnosed with trapeziometacarpal osteoarthritis and healthy subjects will be included in the study. Thickness and cross-sectional area measurements of the thenar muscles of the patient and healthy volunteers will be performed by using Shimadzu SDU 1200-Pro ultrasound system with an 8-10 MHz linear probe. To improve the image quality and to avoid muscle compression, water immersion ultrasonography will be preferred and the hands will be positioned in a water-filled plastic container. The thenar muscles will be imaged in hands of each subject.

In this study, poster-anterior radiographic imaging will be performed. The osteoarthritis stage will be determined on the radiographic image. Three different measurements will be performed on radiography: radial subluxation of the first metacarpal base (RS), articular width (AW) of the first metacarpal, and the distance between the ulnar articular facet of the trapezium and the ulnar edge of the metacarpal (U). RS / AW ratio will be calculated.

Because TMC OA caused pain and affect performance, especially during grip activities in the osteoarthritis and control groups will be tested.

Grip strength will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with trapeziometacarpal osteoarthritis who were between 35 and 75 years

Exclusion Criteria:

* Patient with De'quervain tenosynovitis, trigger finger, entrapment neuropathy and who had undergone hand surgery were excluded.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with trapeziometacarpal osteoarthritis who were between 35 and 75 years and who had the intellectual capacity to give informed consent for the treatment were included in the study.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Ultrasound-based muscle cross-sectional area of thenar muscles in this study will investigate in TMC OA patients and healthy subjects. | through study completion, an average of 1 year
  USG procedures will performed on patients with TMC OA and healthy volunteers. Cross-sectional area measurements of thenar muscles of patient and healthy volunteers will performed using a Shimadzu SDU 1200-Pro ultrasound system with 8-10 MHz linear probe. USG device will calibrated prior to the study. Water bath technique for USG evaluation will preferred in order to improve the image quality and to avoid muscle compression. The hands will positioned in a 60x50x40 cm water-filled plastic container. Five thenar muscles will imaged in the hands of each subject: Opponens pollicis, abductor pollicis brevis, flexor pollicis brevis, first dorsal inteosseous and adductor pollicis muscles. Images will acquired in the cross-sectional planes. 2 evaluators blinded to each other will measure 15 minutes apart. With the first evaluator, it will measure for the second and third times at 30-minute intervals from the first measurement.
Ultrasound-based muscle thickness of thenar muscles in this study will investigate in TMC OA patients and healthy subjects. | through study completion, an average of 1 year
  USG procedures will performed on patients with TMC OA and healthy volunteers.Thickness measurements of thenar muscles of patient and healthy volunteers will performed using a Shimadzu SDU 1200-Pro ultrasound system with 8-10 MHz linear probe. USG device will calibrated prior to the study. Water bath technique for USG evaluation will preferred in order to improve the image quality and to avoid muscle compression. The hands will positioned in a 60x50x40 cm water-filled plastic container. Five thenar muscles will imaged in the hands of each subject: Opponens pollicis, abductor pollicis brevis, flexor pollicis brevis, first dorsal inteosseous and adductor pollicis muscles. Images will acquired in the cross-sectional planes. 2 evaluators blinded to each other will measure 15 minutes apart. With the first evaluator, it will measure for the second and third times at 30-minute intervals from the first measurement.

SECONDARY OUTCOMES:
The radial subluxation rate of the first metacarpal. | through study completion, an average of 1 year
  In this study, while PA radiographic imaging will performed, the elbows will ppositioned in 90 ° flexion, wrists in neutral position, MCP joints at 15-20 ° flexion and nails parallel to each other. During the scanning, patient will toush his thumbs together with maximum force. Three different measurements will made: the radial subluxation (RS) of the first metacarpal base, the articular width of the first metacarpal (AG), and the distance between the ulnar articular facet of the trapezium and the ulnar edge of the metacarpal (U) in milimeter will measured. RS/AG rate will calculated.
Evaluation of functional status of hand | through study completion, an average of 1 year
  Disability of Arm Shoulder and Hand (DASH) will used to determine functional status of hand.The total score is 100, and higher scores indicate a worse functional level.
Grip strength measurement | through study completion, an average of 1 year
  The grip strength will be measured in kilograms using a Jamar Hand Dynamometer
Evaluation of functional status of hand | through study completion, an average of 1 year
  Michigan Hand Outcomes Questionnaire (MHQ) includes 6 subtitles, namely general hand function, ADL, pain, work, aesthetics and satisfaction, and these headings are filled in for theight and left hand. Score calculation for each title is calculated separately. The total score is 100, high scores mean better functional status.
Pain Assessment | through study completion, an average of 1 year
  Pain intensity was evaluated using the visual analog scale (Visual Analogue Scale, VAS). The patients were told that the number "0" means "no pain" and "10" means "unbearable pain" on a 10 cm horizontal line. Patients were asked to mark the severity of pain during rest and activity on this line. The marked place was measured and the result was recorded as the intensity of pain in cm.
Pinch strength measurement | through study completion, an average of 1 year
  The pinch strength will be measured in kilograms using a Pinchmeter.
Minnesota hand skill test | through study completion, an average of 1 year
  Hand skills are evaluated in two different ways, namely placing the discs in their slots and rotating them. People are told that this test is a performance test and they are asked to complete the test as soon as possible. In the insertion part of the test, the patient is asked to take the discs one by one using one hand and put them in the appropriate slots respectively. In the rotating part of the test, the patient is asked to move the discs placed in their nests by rotating the discs in the upper right corner towards the left row. Both tests are repeated 3 times and the result is recorded in seconds.
9 Hole hand skill test | through study completion, an average of 1 year
  This test, which is used to evaluate fine hand skills, is carried out by taking 9 pins from the ground and placing them in the holes and removing them. The test time is approximately 10 minutes. After the patient is told that the test is a performance test and that it will be timed, he is asked to insert the pins first and then remove them as soon as possible. The test is performed twice consecutively on both hands and the two attempts are averaged, the results are recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: ÇİĞDEM AYHAN, ASS. PROF., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Altindağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolf JM, Oren TW, Ferguson B, Williams A, Petersen B. The carpometacarpal stress view radiograph in the evaluation of trapeziometacarpal joint laxity. J Hand Surg Am. 2009 Oct;34(8):1402-6. doi: 10.1016/j.jhsa.2009.06.030. Epub 2009 Sep 10. PMID 19744803
- [Background] Mohseny B, Nijhuis TH, Hundepool CA, Janssen WG, Selles RW, Coert JH. Ultrasonographic quantification of intrinsic hand muscle cross-sectional area; reliability and validity for predicting muscle strength. Arch Phys Med Rehabil. 2015 May;96(5):845-53. doi: 10.1016/j.apmr.2014.11.014. Epub 2014 Dec 4. PMID 25482051
- [Background] Grechenig W, Peicha G, Weiglein A, Tesch P, Lawrence K, Mayr J, Preidler KW. Sonographic evaluation of the thenar compartment musculature. J Ultrasound Med. 2000 Nov;19(11):733-41. doi: 10.7863/jum.2000.19.11.733. PMID 11065261